CLINICAL TRIAL: NCT04940299
Title: A Phase II Study to Assess the Safety and Efficacy of Tocilizumab in Combination With Ipilimumab and Nivolumab in Patients With Advanced Melanoma, Non-Small Cell Lung Cancer, or Urothelial Carcinoma
Brief Title: Tocilizumab, Ipilimumab, and Nivolumab for the Treatment of Advanced Melanoma, Non-Small Cell Lung Cancer, or Urothelial Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1166; NCI-2021-04325 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1166 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-06-18; First posted 2021-06-25 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Locally Advanced Bladder Carcinoma; Locally Advanced Bladder Urothelial Carcinoma; Locally Advanced Lung Non-Small Cell Carcinoma; Locally Advanced Renal Pelvis Carcinoma; Locally Advanced Renal Pelvis Urothelial Carcinoma; Locally Advanced Ureter Urothelial Carcinoma; Locally Advanced Urethral Urothelial Carcinoma; Malignant Solid Neoplasm; Metastatic Bladder Carcinoma; Metastatic Bladder Urothelial Carcinoma; Metastatic Lung Non-Small Cell Carcinoma; Metastatic Melanoma; Metastatic Renal Pelvis Urothelial Carcinoma; Metastatic Ureter Urothelial Carcinoma; Metastatic Urethral Carcinoma; Metastatic Urethral Urothelial Carcinoma; Pathologic Stage III Cutaneous Melanoma AJCC v8; Pathologic Stage IIIA Cutaneous Melanoma AJCC v8; Pathologic Stage IIIB Cutaneous Melanoma AJCC v8; Pathologic Stage IIIC Cutaneous Melanoma AJCC v8; Pathologic Stage IIID Cutaneous Melanoma AJCC v8; Pathologic Stage IV Cutaneous Melanoma AJCC v8; Stage III Bladder Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage III Renal Pelvis Cancer AJCC v8; Stage III Ureter Cancer AJCC v8; Stage III Urethral Cancer AJCC v8; Stage IIIA Bladder Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Bladder Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Bladder Cancer AJCC v8; Stage IV Lung Cancer AJCC v6; Stage IV Renal Pelvis Cancer AJCC v8; Stage IV Ureter Cancer AJCC v8; Stage IV Urethral Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8; Unresectable Melanoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Non-Small-Cell Lung; Melanoma; Urethral Neoplasms; Lung Neoplasms; Ureteral Neoplasms | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab; tocilizumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (ipilimumab, nivolumab, tocilizumab) (Experimental): Patients with melanoma will receive ipilimumab IV over 90 minutes and nivolumab IV over 30 minutes on day 1. Treatment with ipilimumab and nivolumab repeats every 3 weeks for 4 doses, then treatment with nivolumab repeats every 4 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
  Cohort 1 will be divided into 2 sub-groups: sub-group 1 of 25 patients, and subgroup 2 of 10 patients that will consist of varying Tocilizumab administration doses. For sub-group 1, Tocilizumab 162mg will be administered subcutaneously every 2 weeks starting week 0, up to 12 weeks for a total of 6 doses. For sub-group 2 , Tocilizumab 162mg will be administered subcutaneously once every week starting at week 0 up to week 6 followed by Tocilizumab administered subcutaneously every 2 weeks starting at week 6 up to 12 weeks for a total of 9 doses.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab; Biological: Tocilizumab
- Cohort 2 (ipilimumab, nivolumab, tocilizumab) (Experimental): Patients with urothelial cancer will receive ipilimumab IV over 90 minutes and nivolumab IV over 30 minutes on day 1. Treatment with ipilimumab and nivolumab repeats every 3 weeks for 4 doses, then treatment with nivolumab repeats every 4 weeks for 2 years in the absence of disease progression or unacceptable toxicity. Starting on week 1, patients also receive tocilizumab SC every 2 weeks for up to 12 weeks (6 doses) in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab; Biological: Tocilizumab
- Cohort 3 (ipilimumab,, nivolumab, tocilizumab) (Experimental): Patients with NSCLC receive ipilimumab IV over 90 minutes every 6 weeks and nivolumab IV over 30 minutes every 2 weeks for up to 2 years. Patients also receive tocilizumab SC every 2 weeks for up to 12 weeks (6 doses). Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab; Biological: Tocilizumab

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Ipilimumab Biosimilar CS1002; MDX-010; MDX-CTLA4; Yervoy
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
Biological: Tocilizumab — Given SC
  Other Names: Actemra; Immunoglobulin G1, Anti-(Human Interleukin 6 Receptor) (Human-Mouse Monoclonal MRA Heavy Chain), Disulfide with Human-Mouse Monoclonal MRA Kappa-Chain, Dimer; MRA; R-1569; RoActemra

SUMMARY:
This phase II trial investigates the side effects of tocilizumab, ipilimumab, and nivolumab in treating patients with melanoma, non-small cell lung cancer, or urothelial carcinoma that has spread to nearby tissue or lymph nodes (locally advanced). Immunotherapy with monoclonal antibodies, such as ipilimumab and nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Tocilizumab is a monoclonal antibody that may interfere with the immune system to decrease immune-related toxicities. Giving tocilizumab, ipilimumab, and nivolumab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize the safety and tolerability of systemic tocilizumab, an IL-6 receptor antagonist, in combination with Ipilimumab and nivolumab as front-line treatment for patients with advanced cutaneous melanoma, urothelial carcinoma and in EGFR mutant non-small cell lung cancer (NSCLC).

II. To determine the grade 3 or higher toxicity rate of Tocilizumab in combination with Ipilimumab and nivolumab for patients with advanced cutaneous melanoma.

SECONDARY OBJECTIVES:

I. To estimate the objective response rate (ORR), defined as the proportion of patients with complete response (CR) or partial response (PR), and durable response rate (DRR), defined as the proportion of patients with objective responses of > 6 months duration, as determined by Response Evaluation Criteria in Solid Tumors (RECIST 1.1) and immune related RECIST (irRECIST).

II. To estimate progression-free survival (PFS) defined as the time from the start of treatment to disease progression or death, whichever occurs first.

III. To estimate overall survival (OS) defined as the time from the start of treatment to death from any cause.

EXPLORATORY OBJECTIVE:

I. To assess pre- and post-treatment blood/tumor biopsies for immunologic assessment and to explore any potential association between biomarker measurements and antitumor activity.

OUTLINE: OUTLINE: Patients are assigned to 1 of 3 cohorts: 1=melanoma, 2=Urothelial, 3=NSCLC.

COHORT 1: Patients with melanoma will receive ipilimumab intravenously (IV) over 90 minutes and nivolumab IV over 30 minutes on day 1. Treatment with ipilimumab and nivolumab repeats every 3 weeks for 4 doses, then treatment with nivolumab repeats every 4 weeks for 2 years in the absence of disease progression or unacceptable toxicity. Cohort 1 will be divided into 2 sub-groups: sub-group 1 of 25 patients, and subgroup 2 of 10 patients that will consist of varying Tocilizumab administration doses. For sub-group 1, Tocilizumab 162mg will be administered subcutaneously every 2 weeks starting week 0, up to 12 weeks for a total of 6 doses. For sub-group 2 , Tocilizumab 162mg will be administered subcutaneously once every week starting at week 0 up to week 6 followed by Tocilizumab administered subcutaneously every 2 weeks starting at week 6 up to 12 weeks for a total of 9 doses.

COHORT 2: Patients with urothelial cancer will receive ipilimumab IV over 90 minutes and nivolumab IV over 30 minutes on day 1. Treatment with ipilimumab and nivolumab repeats every 3 weeks for 4 doses, then treatment with nivolumab repeats every 4 weeks for 2 years in the absence of disease progression or unacceptable toxicity. Starting on week 1, patients also receive tocilizumab SC every 2 weeks for up to 12 weeks (6 doses) in the absence of disease progression or unacceptable toxicity.

COHORT 3: Patients with NSCLC receive ipilimumab IV over 90 minutes every 6 weeks and nivolumab IV over 30 minutes every 2 weeks for up to 2 years. Patients also receive tocilizumab SC every 2 weeks for up to 12 weeks (6 doses). Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria

1) Signed Written Informed Consent

1. Participants must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal participant care.
2. Participants must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, tumor biopsies, and other requirements of the study.
3. All consented participants should be registered in the institutional database CORe 2) Type of Participant and Target Disease Characteristics

   Cohort 1:

   Melanoma (n=35 patients)
   1. Histologically confirmed stage III (unresectable) or stage IV melanoma, as per American Joint Committee on Cancer (AJCC) Version 8 staging system (Appendix A). Patients must consent to BRAF testing or have documented BRAF status as per regionally acceptable V600 mutational status testing. Specifically, 10 melanoma patients will be initially enrolled, and an additional 25 melanoma patients will be enrolled in expansion cohort. Patients with biopsiable disease will have tissue collected including patients in the expansion cohorts. Archival tumor tissue samples may be collected in place of the biopsy after PI consultation. If biopsy is not feasible, or the patient declines to participate due to the biopsy, the patient may still enroll with PI approval.
   2. Treatment-naïve participants (ie, no prior systemic anticancer therapy for unresectable or metastatic melanoma) with the exception of prior adjuvant treatment for melanoma with approved agents (eg, BRAF/MEK inhibitors, ipilimumab, nivolumab, pembrolizumab or interferon). Participants who have had recurrence within the 6 months of completing adjuvant treatment are not eligible.

   Cohort 2:

   Urothelial Carcinoma (n=10 patients) 1. Histologically or cytologically documented locally advanced or transitional cell carcinoma of the urothelium including renal pelvis, ureters, urinary bladder, or urethra. Patients with mixed histologies are required to have a dominant transitional cell pattern.

   2. Enrollment of urothelial carcinoma 1st line patients who are cisplatin-ineligible and who, after consultation with the investigator, choose to forego front-line chemotherapy or immunotherapy.

   3. Treatment naïve, cisplatin-eligible patients who refuse chemotherapy standard of care or treatment naive, cisplatin-ineligible patients who meet at least one of the following criteria:

   - Common Terminology Criteria for Adverse Events (CTCAE) v5 Grade ≥ 2 audiometric hearing loss. CTCAE v5 Grade ≥ 2 peripheral neuropathy.
   * Cisplatin ineligibility defined as: GFR less than 60 and ≥ 15 mL/min or; CHF NYHA class III or higher or; peripheral neuropathy grade 2 or higher or ECOG PS 2 or higher or; impaired hearing grade 2 or higher.
   * GFR is either measured using a 24 hour urine, calculated using Cockroft-Gault, or estimated using the MDRD method from the National Kidney Disease Education Program (NKDEP) (the method reported by MDACC laboratories).

     a. Cockroft-Gault formula: CLcr = [(140-age) • wt(kg)]/[72 •Creat (mg/dL)] (Multiply by 0.85 for females).

     4. No prior chemotherapy for inoperable locally advanced or metastatic urothelial carcinoma.

     5. Prior local intravesical chemotherapy is allowed if completed at least 4 weeks prior to the initiation of study treatment.

     6. For patients who received prior adjuvant/neoadjuvant chemotherapy or chemo-radiation for urothelial carcinoma, a treatment-free interval of more than 12 months between the last treatment administration and the date of recurrence is required to be considered treatment naive in the metastatic setting. Patients must not have received neoadjuvant or adjuvant therapy with any immuno-oncology regimens. Please note that this small population of patients will be excluded.

   Cohort 3: (n=10 patients)
   1. Subjects diagnosed with histologically or cytologically confirmed locally advanced/metastatic NSCLC with EGFR mutation known to be associated with EGFR TKI sensitivity (including G719X, exon 19 deletion, L858R, L861Q).
   2. Subjects must have received one prior line of therapy with an EGFR TKI in the locally advanced/metastatic setting.
   3. Subjects need to meet either A or B. A) Must have received and progressed on an approved first or second generation EGFR TKI (eg, erlotinib or gefitinib [first generation] or afatinib [second generation]) and must be T790M negative by an approved testing assay on tumor biopsy at the time of progression. B) Patient must have received third generation TKI Osimertinib and progressed on this therapy for study entry. C) TKI needs to be the last therapy. D) Prior chemotherapy received in the neoadjuvant or adjuvant settings will not be considered a line of therapy.

   Common Inclusion Criteria for all three Cohorts

   1. Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1 (adults 18 years or older).

   2. Measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) per RECIST 1.1 criteria.

   3. Participants with stable brain metastases <=3cm, with no clinical requirement for local intervention (surgery, radiosurgery, corticosteroid therapy) or other systemic therapy are allowed to enroll. Subjects must be free of neurologic signs and symptoms related to metastatic intracranial lesions and must not have required or received systemic corticosteroid therapy within 10 days prior to first treatment.

   4. All participants must have tissue submitted during screening. Either a formalin-fixed, paraffin- embedded (FFPE) tissue block or unstained tumor tissue sections, obtained within 3 months prior to enrollment. Biopsy should be excisional, incisional, punch biopsy, core needle or surgical specimen. Fine needle aspiration is unacceptable for submission. Biopsies of bone lesions that do not have a soft tissue component are also unacceptable for submission. If the patient refuses the biopsy, the patient may still enroll with PI approval.

   5. Prior palliative radiotherapy is allowed. Radiation-related toxicities should have resolved to grade 1 or less prior to study entry. Please note that radiated lesions cannot be used as measurable lesions unless there is clear evidence of progression 6. Participants must be able and willing to comply with the study visit schedule and study procedures.

   3) Age and Reproductive Status

<!-- -->

1. Males and females, ages 18 years or older
2. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study treatment.
3. Women must not be breastfeeding
4. Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception for the duration of treatment with study treatment and for 5 months post- treatment completion. Women should use an adequate method(s) of contraception.
5. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study treatment(s) and 7 months post-treatment completion. In addition, male participants must be willing to refrain from sperm donation during this time. Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception.
6. Azoospermic males are exempt from contraceptive requirements. WOCBP who are continuously not heterosexually active are also exempt from contraceptive requirements, and still must undergo pregnancy testing as described in this section.

Investigators shall counsel WOCBP, and male participants who are sexually active with WOCBP, on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise on the use of highly effective methods of contraception, which have a failure rate of < 1% when used consistently and correctly.

Exclusion Criteria

1) Medical Conditions

a) Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity.

b) Uveal melanoma is excluded. c) Any condition including medical, emotional, psychiatric, or logistical that, in the opinion of the Investigator, would preclude the patient from adhering to the protocol or would increase the risk associated with study participation or study drug administration or interfere with the interpretation of safety results (eg, a condition associated with diarrhea or acute diverticulitis).

d) Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.

e) Participants with an active, known or suspected autoimmune disease. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.

f) Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of start of week 0 day 1. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease. Please see Section 4.3for permitted therapies.

g) History of organ transplant or tissue that requires systemic use of immune suppressive agents h) Active infection requiring systemic therapy within 14 days prior to week 0 day 1.

i) Known cardiac history including: i) History of unstable or deteriorating cardiac disease within the previous 12 months prior to screening including but not limited to the following:

(1) Unstable angina or myocardial infarction (2) Transient ischemic attack (TIA)/Cerebrovascular accident (CVA) (3) Congestive heart failure (New York Heart Association [NYHA] Class III or IV) (4) Uncontrolled clinically significant arrhythmias j) Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS). NOTE: Testing for HIV must be performed at sites where mandated locally.

2) Prior/Concomitant Therapy

a) Use of an investigational agent or an investigational device within 28 days before administration of first dose of study drug b) Participants who have received a live / attenuated vaccine within 30 days before first treatment c) Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways with the exception of treatment with adjuvant intent as described in inclusion 2a.

d) Participants with history of life-threatening toxicity related to prior immune therapy (e.g. anti- CTLA-4 or anti-PD-1/PD-L1 treatment or any other antibody or drug specifically targeting T- cell co-stimulation or immune checkpoint pathways) except those that are unlikely to re-occur with standard countermeasures (e.g. Hormone replacement after adrenal crisis) e) Treatment with botanical preparations (eg, herbal supplements or traditional Chinese medicines) intended for general health support or to treat the disease under study within 2 weeks prior to study treatment initiation.

3) Physical and Laboratory Test Findings

1. WBC < 2000/μL
2. Neutrophils < 1500/μL
3. Platelets < 100,000/μL
4. Hemoglobin < 9.0 g/dL NOTE: May not transfuse within 14 days of study treatment initiation to meet eligibility criteria 3a through 3d.
5. Serum creatinine > 1.5 x ULN, unless creatinine clearance ≥ 40 mL/min (measured or calculated using the Cockroft-Gault formula) Female CLcr = (140- age in years) x weight in kg x 0.85 72 x serum creatinine in mg/ dL Male CLcr = (140- age in years) x weight in kg x 1.00 72 x serum creatinine in mg/ dL
6. AST/ALT: > 3.0 x ULN
7. Total bilirubin > 1.5 x ULN (except participants with Gilbert Syndrome who must have a total bilirubin level of < 3.0x ULN)
8. Any positive test result for hepatitis B virus or hepatitis C virus indicating presence of virus, eg, Hepatitis B surface antigen (HBsAg, Australia antigen) positive, or Hepatitis C antibody (anti-HCV) positive (except if HCV-RNA negative).

   4) Allergies and Adverse Drug Reaction

a) History of allergy or hypersensitivity to study drug components b) History of severe hypersensitivity reaction to any monoclonal antibody c) Known hypersensitivity to Tocilizumab, Ipilimumab, or Nivolumab.

5) Other Exclusion Criteria

1. Prisoners or participants who are involuntarily incarcerated. (Note: under certain specific circumstances a person who has been imprisoned may be included or permitted to continue as a participant.
2. Participants who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness

Eligibility criteria for this study have been carefully considered to ensure the safety of the study participants and that the results of the study can be used. It is imperative that participants fully meet all eligibility criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity | Up to 2 years
  Will be summarized overall and for each tumor type using frequencies and percentages.
Occurrence of one or more grade 3 or higher adverse event in a given patient (Cohort 1) | Up to 2 years
  Will be assessed by Common Terminology Criteria for Adverse Events version 5.0. Grade 3 or greater toxicity rate will be computed along with their associated exact 95% confidence interval.

SECONDARY OUTCOMES:
Best overall response | Up to 2 years
  Will be defined by Response Evaluation Criteria in Solid Tumors (RECIST v1.1) and immune related Response Evaluation Criteria in Solid Tumors (irRECIST). Will be computed along with their associated 95% credible interval and exact 95% confidence interval.
Progression-free survival (PFS) | Time from the start of treatment to disease progression (defined by irRECIST) or death, whichever occurs first, assessed up to 2 years
  Will be estimated using the Kaplan-Meier method. Median PFS along with its corresponding 95% confidence intervals will be presented as well as rates at specific timepoints.
Overall survival (OS) | Time from the start of treatment to death from any cause, assessed up to 2 years
  Will be estimated using the Kaplan-Meier method. Median OS along with its corresponding 95% confidence intervals will be presented as well as rates at specific timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Rodabe Amaria, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Fa'ak F, Buni M, Falohun A, Lu H, Song J, Johnson DH, Zobniw CM, Trinh VA, Awiwi MO, Tahon NH, Elsayes KM, Ludford K, Montazari EJ, Chernis J, Dimitrova M, Sandigursky S, Sparks JA, Abu-Shawer O, Rahma O, Thanarajasingam U, Zeman AM, Talukder R, Singh N, Chung SH, Grivas P, Daher M, Abudayyeh A, Osman I, Weber J, Tayar JH, Suarez-Almazor ME, Abdel-Wahab N, Diab A. Selective immune suppression using interleukin-6 receptor inhibitors for management of immune-related adverse events. J Immunother Cancer. 2023 Jun;11(6):e006814. doi: 10.1136/jitc-2023-006814. PMID 37328287
- [Derived] Hailemichael Y, Johnson DH, Abdel-Wahab N, Foo WC, Bentebibel SE, Daher M, Haymaker C, Wani K, Saberian C, Ogata D, Kim ST, Nurieva R, Lazar AJ, Abu-Sbeih H, Fa'ak F, Mathew A, Wang Y, Falohun A, Trinh V, Zobniw C, Spillson C, Burks JK, Awiwi M, Elsayes K, Soto LS, Melendez BD, Davies MA, Wargo J, Curry J, Yee C, Lizee G, Singh S, Sharma P, Allison JP, Hwu P, Ekmekcioglu S, Diab A. Interleukin-6 blockade abrogates immunotherapy toxicity and promotes tumor immunity. Cancer Cell. 2022 May 9;40(5):509-523.e6. doi: 10.1016/j.ccell.2022.04.004. Epub 2022 May 9. PMID 35537412
- See also: MD Anderson Cancer Center — http://www.mdanderson.org